CLINICAL TRIAL: NCT03069664
Title: Palliative Pancreatic Duct Stenting in Patients With Inoperable Pancreatic Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Leena Kylanpaa, MD, PhD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Palliative pancreatic stenting
Record Dates: First submitted 2017-02-19; First posted 2017-03-03 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Pancreatic Cancer; Pancreatic Duct Stricture
Keywords: Pancreatic Cancer; Pancreatic Duct Stricture; Endoscopic treatment
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Covered Self-expandable Metal Stent (Active Comparator): ERCP (endoscopic retrograde cholangiopancreatography) and placement of a pancreatic duct stent
  Interventions: Procedure: ERCP; Device: Covered Self-expandable Metal Stent
- Control group (No Intervention): control group

INTERVENTIONS:
Procedure: ERCP — endoscopic retrograde cholangiopancreatography
  Arms: Covered Self-expandable Metal Stent
Device: Covered Self-expandable Metal Stent — Pancreatic duct stent
  Arms: Covered Self-expandable Metal Stent

SUMMARY:
Patients with pancreatic cancer often suffer from chronic abdominal pain, weight loss and decreased quality of life. The patients also often need pancreatic enzyme supplements. In this prospective study the aim is to see whether patients undergoing palliative pancreatic duct drainage will experience less chronic abdominal pain and a higher quality of life than patients with the same diagnosis without the procedure. The study also investigates whether the nutritional state of the patients with palliative stents remains better than in the control group.

DETAILED DESCRIPTION:
In this prospective study all patients have inoperable pancreatic cancer. In these patients the pancreatic tumor causes radiologically visible dilatation of the pancreatic duct proximally to the tumor with a minimum diameter of 6mm. Patients also suffer from chronic abdominal pain caused by pancreatic cancer. The strength of the pain the patients are experiencing is evaluated with visual analogue scale (VAS). Patients in this study report experiencing chronic abdominal pain at least the strength of VAS 4 at the time of recruitment.

In this pilot study a total of 40 patients are recruited. Patients are divided into to two 20 patient groups. First group will receive a pancreatic duct stent followed by pain medication if needed and the control group will go with conventional pain relief methods only. All patients are asked to evaluate the strength of experienced pain with visual analogue scale at the time of recruitment, and then every 4 weeks up to 24 weeks. The patients will also be asked to evaluate their quality of life with a standardized EORTC-QLQ C30 version 3 quality of life questionnaire at the time of recruitment and then every 4 weeks up to 24 weeks. The patients are also asked to report their body weight, and the amount of pancreatic enzyme supplements needed at every point of survey.

ELIGIBILITY:
Inclusion Criteria:

* Patients have inoperable pancreatic cancer.
* Pancreatic tumor causes radiologically visible dilatation of the pancreatic duct proximally to the tumor with a minimum diameter of 6mm.
* Patients in this study report experiencing chronic abdominal pain at least the strength of VAS 6 (Visual Analogue Scale) at the time of recruitment.

Exclusion Criteria:

* Patients are not fit enough to undergo ERCP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-11-17 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in experienced quality of life | Enquiry at recruitment and every 4 weeks up to 24 weeks
  The patients will be asked to evaluate their quality of life with a standardized EORTC-QLQ C30 version 3 questionnaire at the time of recruitment and then every 4 weeks up to 24 weeks.

SECONDARY OUTCOMES:
Change in experienced strength of pain in visual analogue scale | Enquiry at recruitment and every 4 weeks up to 24 weeks
  Patients evaluate the strength of pain in visual analogue scale
Change in body weight | Enquiry at recruitment and every 4 weeks up to 24 weeks
  Patients report their body weight in kilograms at every point of survey.
Change in need for pancreatic enzyme supplements | Enquiry at recruitment and every 4 weeks up to 24 weeks
  Patients report their need for pancreatic enzyme supplements at every point of survey

CONTACTS AND LOCATIONS:
Overall Officials: Leena Kylänpää, MD, PhD, Principal Investigator — Helsinki UniversityHospital; Sini M Vehviläinen, MD, Study Chair — Helsinki University Central Hospital; Hanna Seppänen, MD, PhD, Study Chair — Helsinki University Central Hospital; Marianne Udd, MD, PhD, Study Chair — Helsinki University Central Hospital; Outi Lindström, MD, PhD, Study Chair — Helsinki University Central Hospital
Locations (2):
- Finland (2):
  - Helsinki University Hospital, Helsinki, HUS
  - Helsinki University Hospital, Helsinki, Uusimaa

IPD SHARING:
Plan to Share IPD: No